CLINICAL TRIAL: NCT00645411
Title: A Combined Phase II/III, Observer-Blind, Randomized, Multi-center Study to Evaluate Safety, Tolerability and Immunogenicity of Trivalent Subunit Influenza Vaccines, Produced Either in Mammalian Cell Culture or in Embryonated Hen Eggs, in Healthy Children and Adolescents
Brief Title: Pediatric Safety and Immunogenicity Study of Cell-Culture Derived and Egg-based Subunit Influenza Vaccines in Healthy Children and Adolescents
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V58P12; Eudract Number: 2007-001534-13
Record Dates: First submitted 2008-03-21; First posted 2008-03-27 (Estimated); Results first posted 2013-01-16 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-10

CONDITIONS: Influenza
Keywords: Influenza; Flu; Cell Culture-Derived; Egg-Derived; Healthy Children; Healthy Adolescents; Safety; Immunogenicity; Trivalent; Inactivated; Vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohorts 1 + Cohort 2 (9-17 Yrs) cTIV (Experimental): All subjects received one 0.5 mL IM injection, of cell culture-derived trivalent influenza vaccine containing 15μg of HA for each strain (A/Solomon Islands/3/2006 [H1N1]-like, A/Wisconsin/67/2005 [H3N2]-like, and B/Malaysia/ 2506/2004-like), recommended for the 2007-2008 influenza season in the Northern Hemisphere
  Interventions: Biological: Cell culture-derived influenza subunit vaccine (cTIV)
- Cohorts 1 + Cohort 2 (9-17 Yrs) eTIV (Active Comparator): All subjects received one 0.5 mL injection, of egg -derived trivalent influenza vaccine containing 15μg of HA for each strain (A/Solomon Islands/3/2006 [H1N1]-like, A/Wisconsin/67/2005 [H3N2]-like and B/Malaysia/ 2506/2004-like), recommended for the 2007-2008 influenza season in the Northern Hemisphere.
  Interventions: Biological: Egg derived influenza subunit vaccine (eTIV)
- Cohort 3 (3-8 Yrs) cTIV (Experimental): All subjects received two 0.5 mL injections, administered four weeks apart, of cell culture-derived trivalent influenza vaccine containing 15μg of HA for each strain (A/Solomon Islands/3/2006 [H1N1]-like, A/Wisconsin/67/2005 [H3N2]-like and B/Malaysia/ 2506/2004-like), recommended for the 2007-2008 influenza season in the Northern Hemisphere
  Interventions: Biological: Cell culture-derived influenza subunit vaccine (cTIV)
- Cohort 3 (3-8 Yrs) eTIV (Active Comparator): All subjects received two 0.5 mL injections, administered four weeks apart of egg -derived trivalent influenza vaccine containing 15μg of HA for each strain (A/Solomon Islands/3/2006 [H1N1]-like, A/Wisconsin/67/2005 [H3N2]-like and B/Malaysia/ 2506/2004-like), recommended for the 2007-2008 influenza season in the Northern Hemisphere
  Interventions: Biological: Egg derived influenza subunit vaccine (eTIV)

INTERVENTIONS:
Biological: Cell culture-derived influenza subunit vaccine (cTIV) — One 0.5 ml injection of the cell culture-derived influenza vaccine in the deltoid muscle, preferably of the nondominant arm.
  Arms: Cohorts 1 + Cohort 2 (9-17 Yrs) cTIV
Biological: Egg derived influenza subunit vaccine (eTIV) — One 0.5 ml injection of the conventional egg-derived influenza vaccine in the deltoid muscle, preferably of the nondominant arm.
  Arms: Cohorts 1 + Cohort 2 (9-17 Yrs) eTIV
Biological: Cell culture-derived influenza subunit vaccine (cTIV) — Two 0.5 mL injections,of the cell culture-derived influenza vaccine in the deltoid muscle, preferably of the nondominant arm, administered four weeks apart.
  Arms: Cohort 3 (3-8 Yrs) cTIV
Biological: Egg derived influenza subunit vaccine (eTIV) — Two 0.5 mL injections of the conventional egg-derived influenza vaccine in the deltoid muscle, preferably of the nondominant arm,administered four weeks apart.
  Arms: Cohort 3 (3-8 Yrs) eTIV

SUMMARY:
The present study is the first study designed to evaluate safety, tolerability and immunogenicity of the cell culture-derived influenza vaccine in healthy children and adolescents aged 3 to 17 years. A step-down approach is utilized in which reactogenicity and safety will be assessed in children and adolescents 9 to 17 years of age (Cohort 1) prior to enrolling additional children and adolescents 9 to 17 years of age (Cohort 2) and children 3 to 8 years of age (Cohort 3).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 9 to 17 years (Cohorts 1 and 2) and 3 to 8 years (Cohort 3), whose parents/legal guardians have given written informed consent prior to study entry. Assent will be obtained from subjects according to age requirements of the ECs/IRBs;
2. In good health as determined by:

   1. medical history,
   2. physical examination,
   3. clinical judgment of the Investigator;
3. Able to comply with all study procedures and available for all clinic visits and telephone calls scheduled in the study.

Exclusion Criteria:

1. Any serious disease, such as:

   1. cancer,
   2. autoimmune disease (including rheumatoid arthritis),
   3. diabetes mellitus,
   4. chronic pulmonary disease,
   5. acute or progressive hepatic disease,
   6. acute or progressive renal disease;
2. History of any anaphylaxis or serious reaction following administration of vaccine, or hypersensitivity to eggs, egg protein, chicken feathers, influenza viral protein, neomycin, polymyxin, or any other vaccine component, chemically related substance, or component of the potential packaging materials;
3. Known or suspected impairment/alteration of immune function, including:

   1. use of immunosuppressive therapy such as systemic corticosteroids known to be associated with the suppression of hypothalamic-pituitary-adrenal (HPA) axis or chronic use of inhaled high-potency corticosteroids within 60 days prior to Visit 1,
   2. cancer chemotherapy,
   3. receipt of immunostimulants within 60 days prior to Visit 1,
   4. receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within 3 months prior to Visit 1 or planned during the full length of the study,
   5. known HIV infection or HIV-related disease;
4. History of Guillain-Barré syndrome;
5. Bleeding diathesis;
6. Surgery planned during the study period;
7. Receipt of another investigational agent within 90 days, or before completion of the safety follow-up period in another study, whichever is longer, prior to enrollment and unwilling to refuse participation in another clinical study through the end of the study;
8. Receipt of another vaccine within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to Visit 1;
9. Laboratory-confirmed influenza disease within 6 months prior to Visit 1;
10. For subjects aged 3 to 8 years old, ever received two doses of an influenza vaccine in one influenza season;
11. Receipt of an influenza vaccine within 6 months prior to Visit 1;
12. Experienced a temperature 38.0°C [100.4°F]) and/or any acute illness within 3 days prior to Visit 1;
13. Pregnant or nursing mother;
14. Female of childbearing potential who is sexually active and has not used acceptable birth control measures for at least 2 months prior to study entry and who does not plan to use acceptable birth control measures during the 3 weeks following vaccination or refuses to have a urine pregnancy test prior to enrollment. Oral, injected, inserted or implanted hormonal contraceptive, diaphragm or condom with spermicidal agent or intrauterine device are considered acceptable forms of birth control;
15. Children of research staff or those living with research staff directly involved with the clinical study. Research staff are individuals with direct study subject contact, indirect contact with study subjects, or study site personnel who have access to any study documents containing subject information. This would include receptionists, persons scheduling appointments or making screening calls, regulatory specialists, laboratory technicians, etc.;
16. Any condition, which in the opinion of the Investigator, might interfere with the evaluation of the study objectives.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3604 (Actual)
Dates: Start 2007-10; Primary Completion 2008-02 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (60):
- United States (16):
  - Site 09, Fayetteville, Arkansas
  - Site 10, Downey, California
  - Site 02, Bardstown, Kentucky
  - Site 14, Metairie, Louisiana
  - Site 01, St Louis, Missouri
  - Site 11, Omaha, Nebraska
  - Site 04, Edison, New Jersey
  - Site 05, Endwell, New York
  - Site 16, Fort Worth, Texas
  - Site 13, San Angelo, Texas
  - Site 12, San Antonio, Texas
  - Site 08, Bountiful, Utah
  - Site 07, Salt Lake City, Utah
  - Site 03, Salt Lake City, Utah
  - Site 06, Burke, Virginia
  - Site 15, Spokane, Washington
- Croatia (9):
  - Site 27:Institute of Public Health, Zagreb, City of Zagreb
  - Site 29: Institute of Public Health, Zagreb, City of Zagreb
  - Site 40:Spec. Pediatric Dispensary, Zagreb, City of Zagreb
  - Site 49: Spec. Pediatric Dispensary, Zagreb, City of Zagreb
  - Site 50: Spec. Pediatric Dispensary, Zagreb, City of Zagreb
  - Site 86: Spec. Pediatric Dispensary, Zagreb, City of Zagreb
  - Site 44:Spec. Pediatric Dispensary, Đakovo, Dakovo
  - Site 43: Spec. Pediatric Dispensary, Sisak, Sisak
  - Site 83, Ljudevita Gaja 2, Djakovo
- Finland (14):
  - Site 70: Espoon rokotetutkimusklinikka, Heikintori, Espoo
  - Site 71: Etelä-Helsingin rokotetutkimusklinikka, Helsinki, Helsinki
  - Site 72: Itä-Helsingin rokotetutkimusklinikka, Helsinki, Helsinki
  - Site 76: Järvenpään rokotetutkimusklinikka, Jarvenpaa, Järvenpää
  - Site 79: Kokkola Vaccine Research Clinic, Rantakatu 7, Kokkola
  - Site 77: Kotkan rokotetutkimusklinikka, Kotka, Kotka
  - Site 78: Kuopio Vaccine Research Clinic, Microkatu 1,Osa/Section A, 3rd Floor Pl1188, Kuopio
  - Site 67: Lahden rokotetutkimusklinikka, Lahti, Lahti
  - Site 75: Oulun rokotetutkimusklinikka, Oulu, Oulu
  - Site 66: Tampereen rokotetutkimusklinikka, Tampere, Pirkanmaa
  - Site 68: Porin rokotetutkimusklinikka, Pori, Pori
  - Site 69: Turun rokotetutkimusklinikka, Turku, Turku
  - Site 73: Itä-Vantaan rokotetutkimusklinikka, Vantaa, Vantaa
  - Site 74: Länsi-Vantaan rokotetutkimusklinikka, Vantaa, Vantaa
- Hungary (8):
  - Site 57: Házi Gyermekorvosi Rendelő, Budapest, Budapest
  - Site 53: Heim Pál Gyermekkórház, Budapest, Budapest
  - Site 52: Ferencvárosi Gyermekorvos Kft., Budapest, Budapest
  - Site 56: Házi Gyermekorvosi Rendelő, Budapest, Budapest
  - Site 54: Házi Gyermekorvosi Rendelő, Budapest, Budapest
  - Site 51: 5053. számú Gyermekorvosi Rendelő, Miskolc, Miskolc
  - Site 55: Revamed kft., Nyíregyháza, Nyíregyháza
  - Site 59: Vas Megyei Markusovszky Lajos, Általános, Rehabilitációs és Gyógyfürdő Kórház, Egyetemi Oktató Kórház, Szombathely, Szombathely
- Italy (5):
  - Site 42: Dipartimento di Medicina Clinica e Sperimentale - Sezione di Igiene e Medicina Preventiva, Ferrara, Ferrara
  - Site 47: Dipartimento Scienze della Salute, Sezione di Igiene e Medicina Preventiva, Univesità di Genova, Genova, Genova
  - Site 41: Ospedale Maggiore della Carità-Clinica Pediatrica, Novara, Novara
  - Site 46: USL 2 Perugia, Distretto del perugino, Centro di Salute n. 4 (Madonna Alta) e n. 6 (Ellera di Corciano del distretto del perugino), Perugia, Perugia
  - Site 45: AUSL 7, Ragusa, Ragusa
- Lithuania (6):
  - Site 35, Kaunas, Kaunas County
  - Site 36, Vilnius, Vilnius County
  - Site 32, Vilnius, Vilnius County
  - Site 34, Vilnius, Vilnius County
  - Site 31, Vilnius, Vilnius County
  - Site 33, Vilnius, Vilnius County
- Romania (2):
  - Site 25, Campulung Muscel, Argeş
  - Site 21, Craiova, Dolj

REFERENCES:
- [Result] Vesikari T, Block SL, Guerra F, Lattanzi M, Holmes S, Izu A, Gaitatzis N, Hilbert AK, Groth N. Immunogenicity, safety and reactogenicity of a mammalian cell-culture-derived influenza vaccine in healthy children and adolescents three to seventeen years of age. Pediatr Infect Dis J. 2012 May;31(5):494-500. doi: 10.1097/INF.0b013e31824bb179. PMID 22301476

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 14 sites in Finland, 16 in the US, 9 in Croatia, 5 in Italy, 6 in Lithuania, 2 in Romania, 8 in Hungary.
Pre-assignment Details: All subjects enrolled were included in the trial.
Groups:
- Cohort 1+2 cTIV (9-17 Years): All subjects aged 9-17 years received one 0.5 mL injection, of Cell Culture-derived trivalent influenza vaccine.
- Cohort 1+2 eTIV (9-17 Years): All subjects aged 9-17 years received one 0.5 mL injection, of egg -derived trivalent influenza vaccine.
- Cohort 3 cTIV (3-8 Years): All subjects aged 3-8 years received two 0.5 mL injections, administered four weeks apart, of Cell Culture-derived trivalent influenza vaccine.
- Cohort 3 eTIV (3-8 Years): All subjects aged 3-8 years received two 0.5 mL injections, administered four weeks apart of egg-derived trivalent influenza vaccine.
Period: Overall Study
Arm/Group | Cohort 1+2 cTIV (9-17 Years) | Cohort 1+2 eTIV (9-17 Years) | Cohort 3 cTIV (3-8 Years) | Cohort 3 eTIV (3-8 Years)
Started | 656 | 318 | 1608 | 1022
Completed | 643 | 312 | 1457 | 919
Not Completed | 13 | 6 | 151 | 103
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 19 | 21
Not completed — Lost to Follow-up | 10 | 5 | 124 | 75
Not completed — Protocol Violation | 1 | 0 | 1 | 0
Not completed — Inappropriate enrollment | 0 | 0 | 4 | 1
Not completed — Unable to classify | 0 | 0 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1+2 eTIV (9-17 Years): All subjects aged 9-17 years received one 0.5 mL injection, of egg-derived trivalent influenza vaccine.
- Total: Total of all reporting groups
Arm/Group | Cohort 1+2 cTIV (9-17 Years) | Cohort 1+2 eTIV (9-17 Years) | Cohort 3 cTIV (3-8 Years) | Cohort 3 eTIV (3-8 Years) | Total
Number analyzed (Participants) | 656 | 318 | 1608 | 1022 | 3604
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.6 (2.6) | 12.6 (2.5) | 5.5 (1.7) | 5.4 (1.7) | 7.4 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 304 | 154 | 795 | 494 | 1747
  Male | 352 | 164 | 813 | 528 | 1857

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers of the Cell Culture-derived Vaccine Compared With the Egg-derived Vaccine in 3 to 8 Year-old Children
Description: To demonstrate non-inferiority of the post vaccination hemagglutination inhibition (HI) geometric mean titer (GMT) of the cell culture-derived influenza (cTIV) vaccine to the corresponding GMT of the egg-derived (eTIV) influenza vaccine, for all three strains, after two injections administered four weeks apart to a subset of children 3 to 8 years of age.
  GMTs were evaluated using two assays, HI egg derived antigen assay and HI cell derived antigen assay.
Time Frame: Day 50 post vaccination
Population: The analysis was performed on the per-protocol dataset
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Cohort 3 eTIV (3-8 Years): All subjects aged 3-8 years received two 0.5 mL injections, administered four weeks apart of egg - derived trivalent influenza vaccine.
Arm/Group | Cohort 3 cTIV (3-8 Years) | Cohort 3 eTIV (3-8 Years)
Number analyzed (Participants) | 524 | 513
Titers
  A/H1N1 (egg derived antigen assay) | 407 [358 to 462] | 477 [419 to 542]
  A/H3N2 (egg derived antigen assay) | 768 [666 to 885] | 1293 [1121 to 1491]
  B (egg derived antigen assay) | 25 [21 to 29] | 44 [38 to 51]
  A/H1N1 (cell derived antigen assay) (N=522,513) | 563 [501 to 634] | 610 [542 to 686]
  A/H3N2 (cell derived antigen assay) (N=522,513) | 858 [744 to 990] | 1329 [1152 to 1533]
  B (cell derived antigen assay) (N=522,513) | 53 [46 to 62] | 62 [53 to 72]
Statistical Analysis 1: Comparison: Cohort 3 cTIV (3-8 Years) vs Cohort 3 eTIV (3-8 Years); Non-inferiority of cTIV to eTIV against A/H1N1 influenza strain as measured by HI egg-derived antigen assay; Test type: Non-Inferiority or Equivalence — Cell derived vaccine was considered non-inferior to egg-derived vaccine in post vaccination HI GMTs if, for all three influenza strains, the lower limit of the two-sided 95% confidence interval (CI) for day 50 ratio of GMTs (cTIV/eTIV) was >0.667; ANOVA; Ratio of GMTs = 0.85, 95% CI 2-sided [0.72 to 1.01]
Statistical Analysis 2: Comparison: Cohort 3 cTIV (3-8 Years) vs Cohort 3 eTIV (3-8 Years); Non-inferiority of cTIV to eTIV against A/H3N2 influenza strain as measured by HI egg-derived antigen assay; Test type: Non-Inferiority or Equivalence — Cell derived vaccine (cTIV ) was considered non-inferior to egg-derived vaccine (eTIV) in postvaccination HI GMTs if, for all three influenza strains, the lower limit of the two-sided 95% confidence interval (CI) for day 50 ratio of GMTs(cTIV/eTIV) was >0.667; ANOVA; Ratio of GMTs = 0.59, 95% CI 2-sided [0.49 to 0.72]
Statistical Analysis 3: Comparison: Cohort 3 cTIV (3-8 Years) vs Cohort 3 eTIV (3-8 Years); Non-inferiority of cTIV to eTIV against influenza B strain as measured by HI egg-derived antigen assay; Test type: Non-Inferiority or Equivalence — Cell derived vaccine (cTIV ) was considered non-inferior to egg-derived vaccine (eTIV)in post vaccination HI GMTs if, for all three influenza strains, the lower limit of the two-sided 95% confidence interval (CI) for day 50 ratio of GMTs (cTIV/eTIV) was >0.667; ANOVA; Ratio of GMTs = 0.56, 95% CI 2-sided [0.46 to 0.68]
Statistical Analysis 4: Comparison: Cohort 3 cTIV (3-8 Years) vs Cohort 3 eTIV (3-8 Years); Non-inferiority of cTIV to eTIV against A/H1N1 influenza strain as measured by HI cell-derived antigen assay; Test type: Non-Inferiority or Equivalence — Cell derived vaccine (cTIV) was considered non-inferior to egg-derived vaccine (eTIV) in post vaccination HI GMTs if, for all three influenza strains, the lower limit of the two-sided 95% confidence interval (CI) for day 50 ratio of GMTs (cTIV/eTIV) was >0.667; ANOVA; Ratio of GMTs = 0.92, 95% CI 2-sided [0.79 to 1.08]
Statistical Analysis 5: Comparison: Cohort 3 cTIV (3-8 Years) vs Cohort 3 eTIV (3-8 Years); Non-inferiority of cTIV to eTIV against A/H3N2 influenza strain as measured by HI cell-derived antigen assay; Test type: Non-Inferiority or Equivalence — Cell derived vaccine (cTIV) was considered non-inferior to egg-derived vaccine (eTIV)in post vaccination HI GMTs if, for all three influenza strains, the lower limit of the two-sided 95% confidence interval (CI) for day 50 ratio of GMTs (cTIV/eTIV) was >0.667; ANOVA; Ratio of GMTs = 0.65, 95% CI 2-sided [0.54 to 0.78]
Statistical Analysis 6: Comparison: Cohort 3 cTIV (3-8 Years) vs Cohort 3 eTIV (3-8 Years); Non-inferiority of cTIV to eTIV against B influenza strain as measured by HI cell-derived antigen assay; Test type: Non-Inferiority or Equivalence — Cell derived vaccine (cTIV) was considered non-inferior to egg-derived vaccine (eTIV)in post vaccination HI GMTs if, for all three influenza strains, the lower limit of the two-sided 95% confidence interval (CI) for day 50 ratio of GMTs (cTIV/eTIV)was >0.667; ANOVA; Ratio of GMTs = 0.87, 95% CI 2-sided [0.71 to 1.06]

2. Primary Outcome: Percentages of Subjects Who Attained Seroconversion or Significant Increase in Antibody Titers in the Cell Culture-derived Vaccine Compared With the Egg-derived Vaccine in 3 to 8 Year-old Children
Description: To demonstrate non-inferiority of the cell culture-derived influenza (cTIV) vaccine to the egg-derived (eTIV) influenza vaccine in the percentage of subjects achieving seroconversion or significant increase in antibody titer post vaccination, for all three strains, after two injections administered four weeks apart in children 3 to 8 years of age.
  Seroconversion rate was evaluated using two assays- HI egg derived antigen assay and HI cell derived antigen assay.
Time Frame: Day 50 post vaccination
Population: The analysis was performed on the per-protocol dataset
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Cohort 3 cTIV (3-8 Years) | Cohort 3 eTIV (3-8 Years)
Number analyzed (Participants) | 524 | 513
Percentages of subjects
  A/H1N1 (egg derived antigen assay) | 94 [92 to 96] | 96 [94 to 97]
  A/H3N2 (egg derived antigen assay) | 77 [73 to 81] | 86 [82 to 89]
  B (egg derived antigen assay) | 38 [34 to 42] | 53 [49 to 58]
  A/H1N1 (cell derived antigen assay) (N=522,513) | 96 [93 to 97] | 96 [94 to 98]
  A/H3N2 (cell derived antigen assay) (N=522,513) | 80 [76 to 83] | 85 [82 to 88]
  B (cell derived antigen assay) (N=522,513) | 58 [54 to 63] | 58 [54 to 63]
Statistical Analysis 1: Comparison: Cohort 3 cTIV (3-8 Years) vs Cohort 3 eTIV (3-8 Years); Non-inferiority of cTIV to eTIV against A/H1N1 influenza strain as measured by HI egg-derived antigen assay; Test type: Non-Inferiority or Equivalence — cTIV was considered non-inferior to eTIV in terms of the percentages of subjects achieving seroconversion or significant increase in antibody titer at day 50 if for all three strains, the lower limit of the two-sided 95% CI around the differences in the percentages of subjects achieving seroconversion and significant increase (cTIV minus eTIV) was >-10%; binomial or the method of Miettinen and; Difference in % (cTIV minus eTIV) = -1, 95% CI 2-sided [-4 to 1]
Statistical Analysis 2: Comparison: Cohort 3 cTIV (3-8 Years) vs Cohort 3 eTIV (3-8 Years); Non-inferiority of cTIV to eTIV against A/H3N2 influenza strain as measured by HI egg-derived antigen assay; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; binomial or Miettinen & Nurimen method; Difference % (cTIV - eTIV) = -9, 95% CI 2-sided [-13 to -4]
Statistical Analysis 3: Comparison: Cohort 3 cTIV (3-8 Years) vs Cohort 3 eTIV (3-8 Years); Non-inferiority of cTIV to eTIV against B influenza strain as measured by HI egg-derived antigen assay; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; binominal or Miettinen &Nurimen method; Difference % (cTIV minus eTIV) = -15, 95% CI 2-sided [-21 to -9]
Statistical Analysis 4: Comparison: Cohort 3 cTIV (3-8 Years) vs Cohort 3 eTIV (3-8 Years); Non-inferiority of cTIV to eTIV against A/H1N1 influenza strain as measured by HI cell-derived antigen assay; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; binominal or Miettinen &Nurimen method; Difference % (cTIV minus eTIV) = -1, 95% CI 2-sided [-3 to 2]
Statistical Analysis 5: Comparison: Cohort 3 cTIV (3-8 Years) vs Cohort 3 eTIV (3-8 Years); Non-inferiority of cTIV to eTIV against A/H3N2 influenza strain as measured by HI cell-derived antigen assay; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; binominal or Miettinen &Nurimen method; Difference % (cTIV minus eTIV) = -5, 95% CI 2-sided [-9.5 to 0]
Statistical Analysis 6: Comparison: Cohort 3 cTIV (3-8 Years) vs Cohort 3 eTIV (3-8 Years); Non-inferiority of cTIV to eTIV against B influenza strain as measured by HI cell-derived antigen assay; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; binominal or Miettinen &Nurimen method; Difference % (cTIV minus eTIV) = 0, 95% CI 2-sided [-6 to 6]

3. Secondary Outcome: Geometric Mean Titers After 1 Dose of the Cell Culture-derived or the Egg-derived Influenza Vaccine in 9 to 17 Year-old Children and Adolescents
Description: To evaluate immunogenicity in terms of Geometric Mean Titers (GMTs) in children 9 to 17 years of age after one injection of either cTIV vaccine or eTIV.
  GMTs were evaluated using two assays, HI egg derived antigen assay and HI cell derived antigen assay.
Time Frame: Day 29 post vaccination
Population: The analysis was performed on the per-protocol dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Cohort 1 cTIV (9-17 Years): All subjects aged 9-17 years received one 0.5 mL injection, of Cell Culture-derived trivalent influenza vaccine
- Cohort 1 eTIV (9-17 Years): All subjects aged 9-17 years received one 0.5 mL injection, of egg-derived trivalent influenza vaccine.
Arm/Group | Cohort 1 cTIV (9-17 Years) | Cohort 1 eTIV (9-17 Years)
Number analyzed (Participants) | 142 | 144
Titers
  Baseline (A/H1N1) egg derived antigen assay | 55 [42 to 72] | 78 [60 to 101]
  Day 29 (A/H1N1) egg derived antigen assay | 879 [728 to 1062] | 1107 [918 to 1334]
  Baseline (A/H3N2) egg derived antigen assay | 121 [94 to 155] | 151 [118 to 193]
  Day 29 (A/H3N2) egg derived antigen assay | 706 [607 to 821] | 1857 [1598 to 2157]
  Baseline (B) Egg derived antigen assay | 9.65 [8.2 to 11] | 9.92 [8.45 to 12]
  Day 29 (B) egg derived antigen assay | 58 [48 to 71] | 105 [86 to 129]
  Baseline(A/H1N1)Cell derived assay | 70 [53 to 92] | 90 [69 to 119]
  Day 29 (A/H1N1) cell derived antigen assay | 1076 [886 to 1307] | 1296 [1069 to 1571]
  Baseline(A/H3N2)cell derived assay(N=141,144) | 125 [98 to 158] | 144 [114 to 182]
  Day 29 (A/H3N2) cell derived antigen assay | 676 [585 to 783] | 1651 [1429 to 1908]
  Baseline(B)cell derived assay(N=141,144) | 22 [18 to 27] | 25 [21 to 30]
  Day 29 (B) cell derived antigen assay | 136 [113 to 163] | 186 [155 to 222]

4. Secondary Outcome: Geometric Mean Ratio After 1 Dose of the Cell Culture-derived or the Egg-derived Influenza Vaccine in 9 to 17 Year-old Children and Adolescents.
Description: Immunogenicity was evaluated in terms of Geometric Mean Ratio (GMRs) in 9 to 17 year-old children and adolescents after one injection of either cTIV vaccine or eTIV.
  The criterion is met according to European (CHMP) guideline if the mean geometric increase GMR (day29/day1) in HI antibody titer is >2.5.
Time Frame: Day 29 post vaccination
Population: The analysis was performed on the per-protocol dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cohort 1 cTIV (9-17 Years) | Cohort 1 eTIV (9-17 Years)
Number analyzed (Participants) | 142 | 144
Ratio
  Day 29 (A/H1N1)egg derived antigen assay | 16 [12 to 21] | 14 [11 to 19]
  Day 29 (A/H3N2) egg derived antigen assay | 5.84 [4.43 to 7.7] | 12 [9.33 to 16]
  Day 29 (B) egg derived antigen assay | 6.03 [4.77 to 7.62] | 11 [8.43 to 13]
  Day29(A/H1N1)cell derived antigen assay(N=141,144) | 15 [12 to 21] | 14 [11 to 19]
  Day29(A/H3N2)cell derived antigen assay(N=141,144) | 5.45 [4.21 to 7.06] | 11 [8.87 to 15]
  Day29(B) cell derived antigen assay(N=141,144) | 6.15 [4.96 to 7.63] | 7.37 [5.96 to 9.12]

5. Secondary Outcome: Percentages of Subjects Who Achieved HI Titers ≥40 After 1 Dose of the Cell Culture-derived Vaccine or the Egg-derived Influenza Vaccine in 9 to 17 Year-old Children and Adolescents
Description: To evaluate immunogenicity in terms of percentage of 9 to 17 year-old children and adolescents achieving HI titers ≥40, after one injection of either the cTIV vaccine or the eTIV vaccine.
  This criterion is met according to European (CHMP) guideline if the percentage of subjects achieving HI titers ≥40 is >70% and according to the US (CBER) guideline is met if the lower bound of the two sided 95%CI for percentage of subjects achieving HI titers ≥40 is ≥70%.
Time Frame: Day 29 post vaccination
Population: The analysis was performed on the per-protocol dataset.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Cohort 1 cTIV (9-17 Years) | Cohort 1 eTIV (9-17 Years)
Number analyzed (Participants) | 142 | 144
Percentages of subjects
  Prevaccination (A/H1N1)egg derived antigen assay | 65 [57 to 73] | 75 [67 to 82]
  Day 29 (A/H1N1) egg derived antigen assay | 99 [96 to 100] | 99 [95 to 100]
  Prevaccination (A/H3N2) egg derived antigen assay | 82 [74 to 88] | 86 [79 to 91]
  Day 29 (A/H3N2) egg derived antigen assay | 100 [97 to 100] | 100 [97 to 100]
  Prevaccination(B)egg derived antigen assay | 17 [11 to 24] | 13 [8 to 19]
  Day 29 (B) egg derived antigen assay | 75 [67 to 82] | 84 [77 to 90]
  Prevaccination (H1N1)cell derived assay(N=141,144) | 67 [59 to 75] | 78 [71 to 85]
  Day 29 (A/H1N1)cell derived antigen assay | 99 [96 to 100] | 98 [94 to 100]
  Prevaccination (H3N2)cell derived assay(N=141,144) | 83 [76 to 89] | 86 [79 to 91]
  Day 29 (A/H3N2) cell derived antigen assay | 100 [97 to 100] | 100 [97 to 100]
  Prevaccination (B) cell derived assay(N=141,144) | 40 [32 to 49] | 47 [38 to 55]
  Day 29 (B) cell derived antigen assay | 95 [90 to 98] | 94 [89 to 98]

6. Secondary Outcome: Percentages of Subjects Who Attained Seroconversion or Significant Increase After 1 Dose of the Cell Culture-derived Vaccine or the Egg-derived Influenza Vaccine in 9 to 17 Year-old Children and Adolescents
Description: Seroconversion or significant increase as per CHMP criteria is defined as percentage of subjects with a pre vaccination HI titer <10 to a post vaccination titer ≥40 or a pre vaccination HI titer ≥10 and a ≥4-fold increase in post vaccination HI antibody titer. According to the CHMP criteria, the percentage of subjects achieving seroconversion or significant increase should be >40%.
  According to the CBER criteria, the lower bound of the two-sided 95% CI for the percentage of subjects achieving seroconversion/significant increase should be ≥40%.
Time Frame: Day 29 post vaccination
Population: The analysis was performed on the per-protocol dataset.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Cohort 1 cTIV (9-17 Years) | Cohort 1 eTIV (9-17 Years)
Number analyzed (Participants) | 142 | 144
Percentages of subjects
  Day 29 (A/H1N1) egg derived antigen assay | 77 [70 to 84] | 77 [69 to 84]
  Day 29 (A/H3N2) egg derived antigen assay | 56 [48 to 65] | 77 [69 to 84]
  Day 29 (B) egg derived antigen assay | 56 [48 to 65] | 71 [63 to 78]
  Day29(A/H1N1)cell derived antigen assay(N=141,144) | 74 [66 to 81] | 74 [66 to 81]
  Day29(A/H3N2)cell derived antigen assay(N=141,144) | 52 [44 to 61] | 78 [70 to 84]
  Day29(B)cell derived antigen assay (N=141,144) | 63 [55 to 71] | 69 [61 to 76]

7. Secondary Outcome: Geometric Mean Titers After Two Doses of the Cell Derived or the Egg Derived Vaccine in 3 to 8 Year-old Children
Description: To evaluate immunogenicity in terms of Geometric Mean Titers (GMTs) in children 3 to 8 years of age after two doses of either cTIV vaccine or eTIV,administered 4 weeks apart.
Time Frame: Day 29 and Day 50 post vaccination
Population: The analysis was performed on the per-protocol dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cohort 3 cTIV (3-8 Years) | Cohort 3 eTIV (3-8 Years)
Number analyzed (Participants) | 524 | 513
Titers
  Baseline (A/H1N1) egg derived antigen assay | 16 [14 to 18] | 15 [13 to 17]
  Day29(A/H1N1)egg derived antigen assay(N=515,507) | 152 [124 to 186] | 157 [128 to 192]
  Day50(A/H1N1)egg derived antigen assay | 407 [358 to 462] | 477 [419 to 542]
  Baseline (A/H3N2) egg derived antigen assay | 68 [58 to 80] | 74 [63 to 87]
  Day29(A/H3N2)egg derived antigen assay(N=515,507) | 584 [478 to 713] | 1075 [880 to 1312]
  Day50(A/H3N2)egg derived antigen assay | 768 [666 to 885] | 1293 [1121 to 1491]
  Baseline (B) egg derived antigen assay | 6.16 [5.86 to 6.48] | 6.24 [5.93 to 6.56]
  Day29(B) egg derived antigen assay (N=515,507) | 19 [16 to 22] | 27 [23 to 33]
  Day 50 (B) egg derived antigen assay | 25 [21 to 29] | 44 [38 to 51]
  Baseline (A/H1N1) cell derived antigen assay | 19 [16 to 22] | 17 [14 to 19]
  Day 29 (A/H1N1) cell derived antigen assay | 234 [194 to 283] | 192 [159 to 232]
  Day50(A/H1N1)cell derived antigen assay(N=522,513) | 563 [501 to 634] | 610 [542 to 686]
  Baseline (A/H3N2) cell derived antigen assay | 75 [64 to 88] | 85 [72 to 99]
  Day 29 (A/H3N2) cell derived antigen assay | 653 [536 to 795] | 1099 [903 to 1339]
  Day50(A/H3N2)cell derived antigen assay(N=522,513) | 858 [744 to 990] | 1329 [1152 to 1533]
  Baseline (B) cell derived antigen assay | 8.22 [7.59 to 8.9] | 8.72 [8.05 to 9.45]
  Day 29 (B) cell derived antigen assay | 29 [24 to 36] | 36 [30 to 44]
  Day50 (B) cell derived antigen assay(N=522,513) | 53 [46 to 62] | 62 [53 to 72]

8. Secondary Outcome: Geometric Mean Ratio After Two Doses of the Cell-derived or the Egg-derived Vaccine in 3 to 8 Year-old Children
Description: To evaluate immunogenicity in terms of Geometric Mean Ratio (GMR) in children 3 to 8 years of age after two doses of either the cTIV vaccine or the eTIV vaccine, administered 4 weeks apart according to the CHMP criteria.
  The criterion is met according to the European (CHMP) guideline if the mean geometric increase (GMR day 29/day 1 and GMR day 50/day 1) in HI antibody titer is >2.5
Time Frame: Day 29 and Day 50 post vaccination
Population: The analysis was performed on the per-protocol dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cohort 3 cTIV (3-8 Years) | Cohort 3 eTIV (3-8 Years)
Number analyzed (Participants) | 524 | 513
Ratio
  Day29 (A/H1N1)egg derived antigen assay(N=515,507) | 9.58 [8.37 to 11] | 11 [9.36 to 12]
  Day 50 (A/H1N1) egg derived antigen assay | 25 [23 to 28] | 33 [29 to 36]
  Day29 (A/H3N2)egg derived antigen assay(N=515,507) | 8.65 [7.4 to 10] | 15 [13 to 17]
  Day 50 (A/H3N2) egg derived antigen assay | 11 [9.84 to 13] | 17 [15 to 20]
  Day 29 (B) egg derived assay (N=515,507 | 3.04 [2.59 to 3.57] | 4.36 [3.71 to 5.12]
  Day 50 (B) egg derived antigen assay | 3.99 [3.49 to 4.57] | 7.04 [6.15 to 8.07]
  Day 29 (A/H1N1) cell derived antigen assay | 13 [11 to 14] | 12 [10 to 13]
  Day50(A/H1N1)cell derived antigen assay(N=522,513 | 30 [27 to 34] | 37 [33 to 42]
  Day 29 (A/H3N2) cell derived antigen assay | 8.73 [7.54 to 10] | 13 [11 to 15]
  Day50(A/H3N2)cell derived antigen assay(N=522,513) | 12 [10 to 13] | 16 [14 to 18]
  Day 29 (B) cell derived antigen assay | 3.59 [3.08 to 4.19] | 4.14 [3.55 to 4.82]
  Day 50 (B) cell derived antigen assay(N=522,513) | 6.5 [5.75 to 7.34] | 7.06 [6.24 to 7.99]

9. Secondary Outcome: Percentages of Subjects Who Achieved HI Titers ≥40 After Two Doses of the Cell Culture Derived or the Egg Derived Influenza Vaccine in 3 to 8 Year-old Children
Description: To evaluate immunogenicity in terms of HI titers ≥40, in children 3-8 years of age after two doses of either cTIV vaccine or eTIV vaccine, administered 4 weeks apart.
  The criterion is met according to European (CHMP) guideline if the percentage of subjects achieving HI titers ≥40 is >70% and according to the US (CBER) guideline if the lower bound of the two sided 95%CI for percentage of subjects achieving HI titers ≥40 is ≥70%.
Time Frame: Day 29 and Day 50 post vaccination
Population: The analysis was performed on the per-protocol dataset.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Cohort 3 cTIV (3-8 Years) | Cohort 3 eTIV (3-8 Years)
Number analyzed (Participants) | 524 | 513
Percentages of subjects
  Prevaccination (A/H1N1) egg derived antigen assay | 35 [30 to 39] | 31 [27 to 35]
  Day29(A/H1N1)egg derived antigen assay (N=515,507) | 72 [68 to 76] | 68 [64 to 72]
  Day 50 (A/H1N1) egg derived antigen assay | 96 [94 to 98] | 97 [95 to 98]
  Prevaccination (A/H3N2) egg derived antigen assay | 67 [62 to 71] | 70 [66 to 74]
  Day29(A/H3N2)egg derived antigen assay(N=515,507) | 87 [84 to 90] | 85 [82 to 88]
  Day50 (A/H3N2) egg derived antigen assay | 96 [94 to 98] | 94 [91 to 96]
  Prevaccination (B) egg derived antigen assay | 4 [3 to 7] | 4 [3 to 6]
  Day 29 (B) egg derived antigen assay (N=515,507) | 35 [30 to 39] | 40 [36 to 45]
  Day 50 (B) egg derived antigen assay | 40 [35 to 44] | 55 [51 to 95]
  Prevaccination (A/H1N1) cell derived antigen assay | 36 [32 to 40] | 33 [29 to 38]
  Day 29 (A/H1N1) cell derived antigen assay | 82 [78 to 85] | 76 [72 to 80]
  Day50(A/H1N1)cell derived antigen assay(N=522,513) | 98 [97 to 99] | 98 [96 to 99]
  Prevaccination (A/H3N2) cell derived antigen assay | 71 [67 to 75] | 75 [71 to 79]
  Day 29 (A/H3N2) cell derived antigen assay | 89 [86 to 92] | 85 [82 to 88]
  Day50(A/H3N2)cell derived antigen assay(N=522,513) | 98 [96 to 99] | 93 [91 to 95]
  Prevaccination (B) cell derived antigen assay | 11 [8 to 14] | 12 [10 to 16]
  Day 29 (B) cell derived antigen assay | 43 [39 to 47] | 45 [40 to 49]
  Day 50 (B) cell derived antigen assay (N=522,513) | 60 [56 to 65] | 62 [57 to 66]

10. Secondary Outcome: Percentages of Subjects Who Achieved Seroconversion or Significant Increase in HI Titers After Two Doses of the Cell Culture-derived Vaccine or the Egg-derived Influenza Vaccine in 3 to 8 Year-old Children
Description: as for outcome 6
Time Frame: Day 29 and Day 50 post vaccination
Population: The analysis was performed on the per-protocol dataset.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Cohort 3 cTIV (3-8 Years) | Cohort 3 eTIV (3-8 Years)
Number analyzed (Participants) | 524 | 513
Percentages of subjects
  Day29(A/H1N1) egg derived antigen assay(N=515,507) | 70 [66 to 74] | 67 [63 to 72]
  Day 50 (H1N1) egg derived antigen assay | 94 [92 to 96] | 96 [94 to 97]
  Day29(A/H3N2) egg derived antigen assay(N=515,507) | 65 [61 to 70] | 78 [74 to 81]
  Day 50 (A/H3N2) egg derived antigen assay | 77 [73 to 81] | 86 [82 to 89]
  Day29(B) egg derived antigen assay(N=515,507) | 33 [29 to 37] | 38 [34 to 43]
  Day 50 (B) egg derived antigen assay | 38 [34 to 42] | 53 [49 to 58]
  Day 29 (A/H1N1) cell derived antigen assay | 79 [75 to 83] | 75 [70 to 78]
  Day50(A/H1N1)cell derived antigen assay(N=522,513) | 96 [93 to 97] | 96 [94 to 98]
  Day 29 (A/H3N2) cell derived antigen assay | 70 [66 to 74] | 76 [72 to 80]
  Day50(A/H3N2)cell derived antigen assay(N=522,513) | 80 [76 to 83] | 85 [82 to 88]
  Day 29 (B) cell derived antigen assay | 40 [36 to 44] | 41 [37 to 45]
  Day 50(B)cell derived antigen assay(N=522,513) | 58 [54 to 63] | 58 [54 to 63]

11. Secondary Outcome: Number of Subjects Reporting Local and Systemic Reactions After 1 Dose of the Cell Culture-derived or the Egg-derived Influenza Vaccine in 9 to 17 Year-old Children and Adolescents.
Description: To evaluate safety and tolerability in terms of number of 9 to 17 year-old children and adolescents (cohorts 1 and 2) reporting local and systemic reactions following of one injection of the cTIV or the eTIV vaccine .
Time Frame: up to 7 days after vaccination
Population: The analysis was performed on the safety dataset
Measure: Number; unit: Subjects
Arm/Group | Cohort 1+2 cTIV (9-17 Years) | Cohort 1+2 eTIV (9-17 Years)
Number analyzed (Participants) | 652 | 316
Subjects
  Any Local | 276 | 141
  Injection site pain | 220 | 120
  Injection site erythema | 91 | 45
  Injection site induration | 44 | 28
  Injection site ecchymosis | 34 | 10
  Injection site swelling | 32 | 17
  Any Systemic | 188 | 95
  Chills | 26 | 13
  Malaise | 60 | 34
  Myalgia | 99 | 59
  Arthralgia | 27 | 17
  Headache | 92 | 44
  Sweating | 14 | 3
  Fatigue | 57 | 41
  Fever (≥38C) (N=651,316) | 5 | 3
  Any Other | 44 | 37
  Stayed at home (n=649,316) | 9 | 10
  Analgesic Medication Used | 42 | 31

12. Secondary Outcome: Number of Subjects Reporting Local and Systemic Reactions After One and Two Doses of the Cell Culture-derived Vaccine or Egg-derived Influenza Vaccine in 3 to 8 Year-old Children.
Description: To evaluate the safety and tolerability of the cTIV and the eTIV influenza vaccines in 3 to 8 year-old children terms of number of participants reporting local and systemic reactions after each vaccination.
Time Frame: up to 7 days after each vaccination
Population: The analysis was performed on the safety dataset set.
Measure: Number; unit: Subjects
Groups:
- Cohort 3 eTIV (3-8 Years): All subjects aged 3-8 years received two 0.5 mL injections, administered four weeks apart of egg- derived trivalent influenza vaccine.
Arm/Group | Cohort 3 cTIV (3-8 Years) | Cohort 3 eTIV (3-8 Years)
Number analyzed (Participants) | 1599 | 1013
Subjects
  Injection site pain | 653 | 398
  Injection site erythema | 337 | 206
  Injection site induration | 141 | 84
  Injection site ecchymosis | 144 | 99
  Injection site swelling | 119 | 85
  Chills | 70 | 68
  Malaise | 156 | 117
  Myalgia | 202 | 119
  Arthralgia | 65 | 28
  Headache | 182 | 144
  Sweating | 47 | 28
  Fatigue | 210 | 170
  Fever (≥ 38C) | 75 | 60
  Oral temp; 38 to <38.9 C (N=1598,1013) | 48 | 43
  Stayed at home (N=1582,1003,1519, 955) | 77 | 63
  Analgesic Medication Used | 221 | 148
  Oral temp; 39 to < 40 C (N=1598,1013) | 16 | 15
  Oral temp; ≥ 40 C (N=1598,1013) | 6 | 1

ADVERSE EVENTS:
Time Frame: Throughout the study period (Day 1-181 for Cohorts 1 and 2, and Day 1-209 for cohort 3)
Description: Solicited AEs - day 1 through day 7 after vaccination. All AEs- day 1 through day 29 ( cohort 1&2); day 1 through day 50 (cohort 3). SAEs, onset of chronic illness, and AEs that lead to withdrawal from the study and associated concomitant medications-day 29 to day 181 (cohort 1&2); day 50 through day 209 (cohort 3)
Groups:
- Cohort 3 cTIV (3-8 Yrs; 1st Vaccination); Cohort 3 cTIV (3-8 Yrs; 2nd Vaccination): All subjects aged 3-8 years received two 0.5 mL injections, administered four weeks apart, of Cell Culture-derived trivalent influenza vaccine.
- Cohort 3 eTIV (3-8 Yrs; 1st Vaccination); Cohort 3 eTIV (3-8 Yrs; 2nd Vaccination): All subjects aged 3-8 years received two 0.5 mL injections, administered four weeks apart of egg-derived trivalent influenza vaccine.
Arm/Group | Cohort 1+2 cTIV (9-17 Years) | Cohort 1+2 eTIV (9-17 Years) | Cohort 3 cTIV (3-8 Yrs; 1st Vaccination) | Cohort 3 eTIV (3-8 Yrs; 1st Vaccination) | Cohort 3 cTIV (3-8 Yrs; 2nd Vaccination) | Cohort 3 eTIV (3-8 Yrs; 2nd Vaccination)
Serious Adverse Events (participants affected / at risk) | 5/652 | 3/316 | 2/1599 | 0/1013 | 7/1557 | 5/977
Other Adverse Events (participants affected / at risk) | 328/652 | 168/316 | 799/1599 | 507/1013 | 670/1557 | 413/977
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1+2 cTIV (9-17 Years) (N=652) | Cohort 1+2 eTIV (9-17 Years) (N=316) | Cohort 3 cTIV (3-8 Yrs; 1st Vaccination) (N=1599) | Cohort 3 eTIV (3-8 Yrs; 1st Vaccination) (N=1013) | Cohort 3 cTIV (3-8 Yrs; 2nd Vaccination) (N=1557) | Cohort 3 eTIV (3-8 Yrs; 2nd Vaccination) (N=977)
Thalassemia beta (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendix disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroentritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body height below normal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1+2 cTIV (9-17 Years) (N=652) | Cohort 1+2 eTIV (9-17 Years) (N=316) | Cohort 3 cTIV (3-8 Yrs; 1st Vaccination) (N=1599) | Cohort 3 eTIV (3-8 Yrs; 1st Vaccination) (N=1013) | Cohort 3 cTIV (3-8 Yrs; 2nd Vaccination) (N=1557) | Cohort 3 eTIV (3-8 Yrs; 2nd Vaccination) (N=977)
Fatigue (General disorders) | 57 (67) | 41 (47) | 155 (171) | 119 (143) | 99 (110) | 82 (92)
Injection site erythema (General disorders) | 91 (94) | 45 (45) | 197 (198) | 138 (139) | 209 (211) | 118 (121)
Injection site induration (General disorders) | 44 (44) | 28 (29) | 87 (89) | 44 (45) | 66 (66) | 51 (51)
Injection site pain (General disorders) | 220 (227) | 120 (122) | 451 (462) | 251 (261) | 421 (430) | 266 (278)
Injection site haemorrhage (General disorders) | 34 (37) | 10 (11) | 98 (106) | 60 (67) | 52 (58) | 43 (51)
Malaise (General disorders) | 60 (68) | 34 (41) | 103 (118) | 78 (85) | 76 (86) | 50 (56)
Pyrexia (General disorders) | 12 (13) | 5 (7) | 88 (96) | 73 (84) | 63 (70) | 44 (49)
Myalgia (Musculoskeletal and connective tissue disorders) | 99 (107) | 59 (67) | 141 (150) | 76 (88) | 100 (103) | 67 (70)
Headache (Nervous system disorders) | 99 (125) | 47 (56) | 143 (167) | 111 (135) | 94 (110) | 73 (89)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 4 (4) | 124 (130) | 75 (87) | 70 (75) | 51 (52)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days